CLINICAL TRIAL: NCT03270618
Title: Accuracy Evaluation of A CAD/CAM Surgical Template for Mandible Distraction
Brief Title: Accuracy of a CAD/CAM Surgical Template for Mandible Distraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Xudong Wang, Director of the Department of Oral and Craniomaxillofacial Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cmfs02
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Facial Asymmetry; Mandible; Hypoplasia, Unilateral Condylar; Distraction of Bone
MeSH Terms: conditions — Facial Asymmetry; Diastasis, Bone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CAD/CAM Surgical Template — The templates were designed based on virtual planning and manufactured using three-dimensional printing technique. The template is designed to assist the surgeon to perform the osteotomy and predrill the screw holes to guide the distractor position.

SUMMARY:
The purpose was to assess the accuracy and clinical validation of virtual planning and surgical template in mandible distraction osteogenesis. Patients with hemifacial microsomia were enrolled. Virtual planning and simulation were performed on three-dimensional models. Distraction was simulated on virtual model and the new morphology of the mandible was predicted. The position and direction of the distractor was determined to achieve the optimal morphology. The templates were designed based on virtual planning and manufactured using three-dimensional printing technique. The template is designed to assist the surgeon to perform the osteotomy and predrill the screw holes to guide the distractor position. The outcome evaluation was completed by comparing planned outcomes with postoperative outcomes. Linear and angular differences for the distractor was measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled to undergo mandibular DO via intraoral approach
* Patients who were scheduled to undergo CT scan as a part of their diagnosis and treatment
* Patients who agreed to participate in this study

Exclusion Criteria:

* Patients requiring more than one distractor of the mandible
* Patients with mandible defect
* Patients with previous mandibular trauma

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Linear differences of the distractor position | within latency period (5-7 days after the surgery)
angular differences of the distractor vector | within latency period (5-7 days after the surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Wang, Study Chair — Ninth People's Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No